CLINICAL TRIAL: NCT05082181
Title: NYU Managing Epilepsy Well (MEW) Study: A Randomized Controlled Trial of Telephone-Based Support for People With Epilepsy
Brief Title: Telephone-Based Support Programs for People With Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-00446
Record Dates: First submitted 2021-09-30; First posted 2021-10-18 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy
Keywords: Epilepsy; Depression; Seizures; Quality of life; Mindfulness; Telehealth
MeSH Terms: conditions — Epilepsy; Depression; Seizures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: UPLIFT (Using Practice and Learning to Increase Favorable Thoughts) (Experimental): UPLIFT is a telephone-based depression self-management program for people with epilepsy.
  Interventions: Behavioral: UPLIFT (Using Practice and Learning to Increase Favorable Thoughts)
- Arm 2: BOOST (Bringing Out Our Strength Together) (Active Comparator): BOOST is a telephone-based support program for people with epilepsy.
  Interventions: Behavioral: BOOST (Bringing Out Our Strength Together)

INTERVENTIONS:
Behavioral: UPLIFT (Using Practice and Learning to Increase Favorable Thoughts) — UPLIFT is an 8-week program that combines cognitive behavioral therapy (CBT) and mindfulness techniques and is delivered to small groups of participants by phone. Each weekly session is 1 hour long and is comprised of a check-in period, teaching on the week's topic, group discussion, a skill-building exercise, and a home practice assignment. CBT-related skills include thought monitoring, identifying cognitive distortions, problem identification, goal setting, and identifying supports. Relaxation exercises are also used for coping and to facilitate awareness of the body. Mindfulness activities include attention to breath, sights and sounds and other meditations. Audio guides are provided for home practice of mindfulness exercises.
  Arms: Arm 1: UPLIFT (Using Practice and Learning to Increase Favorable Thoughts)
Behavioral: BOOST (Bringing Out Our Strength Together) — BOOST is a telephone-based support program delivered in 8 weekly group sessions. Each weekly session is 1 hour long and is comprised of a check-in period, introduction of the week's topic, and group discussion. Weekly BOOST session topics include: (1) personal experience of epilepsy; (2) personal experience of mood problems (depression, anxiety, stress); (3) seizure triggers; (4) concerns related to epilepsy treatment (e.g., medication adherence, side effects); (5) changes in seizures over time; (6) the impact of behavior (e.g., sleep, substance use) on seizures; (7) social relationships and epilepsy; and (8) review of the BOOST experience.
  Arms: Arm 2: BOOST (Bringing Out Our Strength Together)

SUMMARY:
This is a two-arm randomized controlled trial to compare telephone-based depression self-management (UPLIFT) to telephone-based support groups (BOOST). A sample of 120 English- and Spanish-speaking people with epilepsy (PWE) with elevated depressive symptoms will be enrolled. Both interventions are 8-week programs delivered in one-hour weekly sessions to groups of about 6 participants. Changes in depressive symptoms, quality of life and seizures will be assessed over 12 months. The trial will also examine mediators and moderators of treatment effects.

DETAILED DESCRIPTION:
The objectives of the trial are:

1. To test effects of UPLIFT versus BOOST on changes in depressive symptoms (primary outcome) in PWE over 12 months.
2. To test effects of UPLIFT versus BOOST on changes in quality of life and seizures (secondary outcomes) in PWE over 12 months.
3. To test whether intervention effects are mediated by increases in mindfulness and decreases in rumination.
4. To test whether intervention effects are moderated by participant characteristics and facilitator characteristics.

ELIGIBILITY:
Inclusion Criteria:

* adult (≥18 years of age);
* diagnosed with epilepsy for at least one year;
* fluent in English or Spanish;
* elevated depressive symptoms (PHQ-9 score ≥10);
* willing to participate in audiotaped group telephone sessions

Exclusion Criteria:

* severe depressive symptoms (PHQ-9 ≥20);
* active suicidal ideation (PHQ-9 item #9 ≥1 or otherwise reported during screening);
* active psychotic disorder (psychiatric diagnosis or antipsychotic medications in the EHR);
* significant cognitive impairment (indicated in EHR or evident during screening)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Presence of clinically significant depressive symptoms | Baseline Visit
  The primary outcome is a dichotomous measure of depressive symptoms based on a Patient Health Questionnaire (PHQ-9) score of <5 versus ≥5. The PHQ-9 assesses depressive symptoms in the past two weeks. Total scores range from 0-27 with recommended cutoffs for mild (5-9), moderate (10-14), moderately severe (15-19) and severe (≥20) depressive symptoms. A PHQ-9 score of <5 indicates absence of clinically significant depressive symptoms.
Presence of clinically significant depressive symptoms | 3 month visit
  The primary outcome is a dichotomous measure of depressive symptoms based on a Patient Health Questionnaire (PHQ-9) score of <5 versus ≥5. The PHQ-9 assesses depressive symptoms in the past two weeks. Total scores range from 0-27 with recommended cutoffs for mild (5-9), moderate (10-14), moderately severe (15-19) and severe (≥20) depressive symptoms. A PHQ-9 score of <5 indicates absence of clinically significant depressive symptoms.
Presence of clinically significant depressive symptoms | 6 month visit
  The primary outcome is a dichotomous measure of depressive symptoms based on a Patient Health Questionnaire (PHQ-9) score of <5 versus ≥5. The PHQ-9 assesses depressive symptoms in the past two weeks. Total scores range from 0-27 with recommended cutoffs for mild (5-9), moderate (10-14), moderately severe (15-19) and severe (≥20) depressive symptoms. A PHQ-9 score of <5 indicates absence of clinically significant depressive symptoms.
Presence of clinically significant depressive symptoms | 12 month visit
  The primary outcome is a dichotomous measure of depressive symptoms based on a Patient Health Questionnaire (PHQ-9) score of <5 versus ≥5. The PHQ-9 assesses depressive symptoms in the past two weeks. Total scores range from 0-27 with recommended cutoffs for mild (5-9), moderate (10-14), moderately severe (15-19) and severe (≥20) depressive symptoms. A PHQ-9 score of <5 indicates absence of clinically significant depressive symptoms.

SECONDARY OUTCOMES:
Change in depressive symptom severity | Baseline Visit, 3 month visit, 6 month visit, 12 month visit
  Continuous PHQ-9 scores will be used to evaluate the magnitude of change in depressive symptoms. The PHQ-9 consists of nine questions that ask respondents how often they've "been bothered by any of the following problems" in the past two weeks. The questions address sleep, energy, appetite, and other possible symptoms of depression. Scores are calculated based on how frequently a person experiences these feelings. Score of 1-4 is considered minimal depression; score of 5-9 is considered mild depression; score of 10-14 is considered moderate depression; score of 15-19 is considered moderately severe depression; score of 20-27 is considered severe depression.
Change in seizure frequency | Baseline Visit, 3 month visit, 6 month visit, 12 month visit
  This will be assessed by self-reported 30-day seizure counts.
Change in seizure severity | Baseline Visit, 3 month visit, 6 month visit, 12 month visit
  This will be assessed by a 12-item version of the Liverpool Seizure Severity Scale. The possible scoring ranges are between 7 and 32 for the percept scale and between 10 and 48 for the ictal/postictal scale. The higher the score the more severe the seizures.
Change in disease-specific quality of life | Baseline Visit, 3 month visit, 6 month visit, 12 month visit
  This will be assessed by the Quality of Life in Epilepsy-10 (QOLIE-10) questionnaire, a 10-item measure of epilepsy-specific aspects of qualify of life. The QOLIE-10-P is a brief survey of health-related quality of life for adults with epilepsy. There are 10 questions about health and daily activities, one question about how much distress you feel about problems and worries related to epilepsy, and a review of what bothers you most.
Change in general health-related quality of life | Baseline Visit, 3 month visit, 6 month visit, 12 month visit
  This will be assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS-10) questionnaire, a 10-item measure of global health (physical, mental and social functioning) developed by NIH as an indicator for Healthy People 2020. The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.

OTHER OUTCOMES:
Change in perceived social support | Baseline Visit, 3 month visit, 6 month visit, 12 month visit
  This will be assessed by the Interpersonal Support Evaluation List, a 12-item measure of the perceived availability of social support resources (appraisal, belonging, tangible support). The ISEL-12 can be scored by summing the items to create an overall social support score; three subscale scores representing appraisal, belonging, and tangible social support have also been proposed.
Change in mindfulness | Baseline Visit, 3 month visit, 6 month visit, 12 month visit
  This will be assessed by the Five Facet Mindfulness Questionnaire Short Form, a 15-item measure that assesses five dimensions of trait mindfulness: observing, describing, acting with awareness, non-judging of inner experience and non-reactivity to inner experience. The following is the scoring information: Observing items: 1, 6, 11; Describe items: 2, 7R, 12 ; Acting with awareness items: 3R, 8R, 13R ; Non-judging items: 4R, 9R, 14R; Non-reactivity items: 5, 10, 15.
Change in rumination | Baseline Visit, 3 month visit, 6 month visit, 12 month visit
  This will be assessed by the Ruminative Responses Scale, a 22-item measure that assesses how often participants engage in ruminative behaviors and cognitions in response to feeling sad or depressed.Each item are rated on a 4-point Likert scale ranging from 1 (never) to 4 (always). The total score ranges from 22 to 88, with higher scores indicating higher degrees of ruminative symptoms.
Change in perceived stress | Baseline Visit, 3 month visit, 6 month visit, 12 month visit
  This will be assessed by the Perceived Stress Scale, a 10-item measure of the degree which situations in one's life are appraised as overwhelming, uncontrollable and unpredictable over the last month. The Perceived Stress Scale (PSS) is a classic stress assessment instrument. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Change in anxiety | Baseline Visit, 3 month visit, 6 month visit, 12 month visit
  This will be assessed by the Generalized Anxiety Disorder-7 Scale, a 7-item measure of anxiety symptoms in the past two weeks that is used to screen for clinically significant anxiety. This is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21. The higher the score, the greater the anxiety
Change in epilepsy self management | Baseline Visit, 3 month visit, 6 month visit, 12 month visit
  This will be assessed by the Epilepsy Self-Management Scale, a 38-item measure of the frequency of use of epilepsy self-management behaviors. The ESMS scores range from 38 to 190, with higher scores reflecting an increased utilization of epilepsy self-management techniques.
Change in self-compassion | Baseline Visit, 3 month visit, 6 month visit, 12 month visit
  This will be assessed by the Self-Compassion Scale, a 12-item measure of thoughts, emotions and behaviors associated with self-compassion. Average overall self-compassion scores tend to be around 3.0 on the 1-5 scale, a score of 1-2.5 indicates low self-compassion, 2.5-3.5 indicates moderate self-compassion and 3.5-5.0 means high self compassion.
Change in healthcare utilization | Baseline Visit, 3 month visit, 6 month visit, 12 month visit
  Self-reported outpatient (neurology/epilepsy and primary care/other specialist) and inpatient encounters will be obtained at each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Spruill, Principal Investigator — NYU Langone Health; Daniel Friedman, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to Tanya.Spruill@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.